CLINICAL TRIAL: NCT02407574
Title: Assessment of the Force Frequency Relationship of the Myocardium After On-pump CABG Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Professor, Head of Department, University of Liege
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FFR2015
Record Dates: First submitted 2015-03-24; First posted 2015-04-03 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Adult Cardiac Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spontaneous rhythm first (Experimental): Stepwise preload increase by repeated administration of 100 mL of fluid during spontaneous rhythm and then stepwise preload reduction by repeated drainage of 100 mL of fluid during atrial pacing.
  Interventions: Device: External Pacing Box
- Atrial pacing first (Experimental): Stepwise preload increase by repeated administration of 100 mL of fluid during atrial pacing and then stepwise preload reduction by repeated drainage of 100 mL of fluid during spontaneous rhythm.
  Interventions: Device: External Pacing Box

INTERVENTIONS:
Device: External Pacing Box — Atrial pacing using an external pacing box

SUMMARY:
The aim of the study is to determine whether increasing the heart rate by epicardial atrial pacing after surgery improves the contractile force of the myocardium. After complete weaning from CPB, several pressure-loops of the LV will be recorded at different levels of preload using transoesophageal echo, invasive blood pressure monitoring. The preload will be manipulated by adding fluid from the CPB reservoir or draining fluid into the CPB reservoir.

ELIGIBILITY:
Inclusion Criteria:

* CABG only surgery
* Preopeartive LVEF ≥ 53 %
* Use of epicardial pacing wires to assist CPB weaning

Exclusion Criteria:

* Contra-indication to TEE
* AV block at the time of CPB weaning
* Sinus rhythm less than 50 or more than 90 BPM after CPB weaning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
End-systolic elastane of the left ventricle. | 30 minutes after CPB weaning